CLINICAL TRIAL: NCT05787548
Title: Reducing Emergency Department Utilization With an After Visit Summary Nudge Toward Alternative Care Options
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0340
Record Dates: First submitted 2023-03-08; First posted 2023-03-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Behavior, Health
Keywords: Emergency Department Use; Urgent Care Use
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard practice (No Intervention): Patients in this arm will receive the current standard practice AVS.
- Contact us first (Experimental): Patients in this arm will receive the standard AVS, plus information on how to contact Geisinger if they need medical attention.
  Interventions: Behavioral: Contact information
- Contact us first + urgent care map (Experimental): Patients in this arm will receive the standard AVS, plus information on how to contact Geisinger if they need medical attention, plus a map to their nearest Geisinger urgent care location and additional information about urgent care.
  Interventions: Behavioral: Contact information; Behavioral: Urgent care map
- Contact us first + urgent care map + self-triage (Experimental): Patients in this arm will receive the standard AVS, plus information on how to contact Geisinger if they need medical attention, plus a map to their nearest Geisinger urgent care location and additional information about urgent care. This arm will also receive a self-triage chart, with common reasons patients go to the ED and situations where seeking alternative care might be appropriate.
  Interventions: Behavioral: Contact information; Behavioral: Urgent care map; Behavioral: Self-triage chart

INTERVENTIONS:
Behavioral: Contact information — Information on how to contact Geisinger if the patient needs care
  Arms: Contact us first; Contact us first + urgent care map; Contact us first + urgent care map + self-triage
Behavioral: Urgent care map — A map of the patient's nearest Geisinger urgent care location, with information about urgent care
  Arms: Contact us first + urgent care map; Contact us first + urgent care map + self-triage
Behavioral: Self-triage chart — A chart demonstrating what to do in response to several common conditions where the patient might be compelled to visit the ED
  Arms: Contact us first + urgent care map + self-triage

SUMMARY:
Decreasing utilization of the Emergency Department (ED) is a priority for the system. Often, ED visits can be avoided if patients contact Geisinger first to get appropriate direction for their concern or are otherwise better informed about reasons to visit the ED vs. urgent care or primary care facilities. The study team is working to reduce ED utilization by including additional information in adult outpatient After Visit Summaries (AVSs). The study will involve will involve A/B testing different AVS versions, including 1) a version that encourages patients to contact Geisinger via different contact methods, 2) a version that includes a map to the patient's closest ConvenientCare location and accompanying information about ConvenientCare, and 3) a version that includes a self-triage guide. A control group will receive the current standard AVS. Analysis results will be assessed to determine which version is most effective at reducing ED use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Has a Geisinger Primary Care Physician assigned
* Completes an outpatient office visit or telemedicine appointment at Geisinger

Exclusion Criteria:

* The AVS was not printed according to the EHR, and the patient does not have an active MyGeisinger patient portal account, so they do not have a way to view the AVS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239841 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Inappropriate ED visits | In the 30 days following the appointment
  Visited the ED inappropriately (y/n)
  We will apply the NYU algorithm (Ballard et al., 2010) to determine whether an ED visit is inappropriate.

OTHER OUTCOMES:
Urgent care visits | In the 30 days following the appointment
  Visited urgent care (y/n)
Calls | In the 30 days following the appointment
  Called Geisinger (y/n)
Patient portal messages | In the 30 days following the appointment
  Sent a patient portal message (y/n)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT05787548/Prot_SAP_001.pdf